CLINICAL TRIAL: NCT02460341
Title: The Effects of Ondansetron on Brain Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Emily Stern, Assistant Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: GCO 14-1794
Record Dates: First submitted 2015-05-28; First posted 2015-06-02 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Brain Function; Healthy Adults
Keywords: fMRI; Brain function; Sensory processing
MeSH Terms: interventions — Ondansetron

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ondansetron-8 (Experimental): Single dose of 8 mg ondansetron (crossover with single dose of placebo)
  Interventions: Drug: ondansetron; Drug: placebo
- ondansetron-16 (Experimental): Single dose of 16 mg ondansetron (crossover with single dose of placebo)
  Interventions: Drug: ondansetron; Drug: placebo
- ondansetron-24 (Experimental): Single dose of 24 mg ondansetron (crossover with single dose of placebo)
  Interventions: Drug: ondansetron; Drug: placebo

INTERVENTIONS:
Drug: ondansetron — Ondansetron 8mg, 16mg, 24mg
  Other Names: Zofran
Drug: placebo — placebo pill

SUMMARY:
This project investigates the effects of a single dose of ondansetron on brain function in healthy adults. The investigators hypothesize that there will be a dose-dependent reduction in activation of the insula and somatosensory brain regions associated with the use of ondansetron.

DETAILED DESCRIPTION:
Objectives:

The overall objective of this study is to examine the effects of single doses of 8 mg, 16 mg, and 24 mg ondansetron as compared to placebo on neural mechanisms of cognition and perception in healthy individuals.

Background:

Many psychiatric disorders are associated with altered sensory experiences arising from within the body. Examples include increased experience of sensations or urges in muscles, skins, joints or visceral organs in tic disorders, OCD patients with symptoms of "not just right experiences" or disgust sensitivity, and impulse control disorders (ICDs) such as trichotillomania or skin-picking. In OCD, sensory phenomena occur in approximately half of patients, are associated with earlier age of onset, and may be harder to treat with classic cognitive-behavioral approaches to OCD. Of interest, sensory phenomena in OCD are associated with Tourette's syndrome and respond to pharmacological treatments primarily used for tics. As such, abnormal sensory processing may be a basic mechanism that links various psychiatric disorders.

The process of attending to body sensations is referred to as interoception, and broadly includes the detection of, or attention to, experiences arising from the viscera and soma. Research has revealed a cortical interoceptive circuit involving insula, anterior cingulate cortex (ACC), and somatomotor cortex.

Ondansetron (OND) is a good candidate for the modulation of the above-described interoceptive circuit. It is a selective 5-HT3 (serotonin) receptor antagonist that acts on both peripheral and central receptors. OND has long been used to treat nausea and vomiting due to chemotherapy, radiation therapy, anesthesia, and opioid-induced emesis. It has also been used alone or as adjunctive therapy for the treatment of both OCD and Tourette's disorder, showing some efficacy in small clinical trials. The mechanisms by which ondansetron improves symptoms in OCD and tic disorders are unknown, but a recent study found that OND application directly into the insula decreased disgust reactions in rats. This data suggests that ondansetron's clinical efficacy could be related to effects on interoceptive circuit activity in the insula and sensorimotor regions, a possibility that is being explored in the current protocol. Typical dosages for anti-emetic action is 8-24 mg. The investigator's pilot data found that a single 16 mg dose of ondansetron reduced activation of insula and somatosensory cortex in both healthy controls and patients with OCD. As a follow-up to this pilot work, the current protocol will compare the effects of three different dosages of ondansetron (8 mg, 16 mg, and 24 mg) on activation in insula and somatosensory cortex during tasks of cognition and perception in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* All subjects must be medically healthy, between 18 and 60 years of age, and fluent (speaking and writing) in English

Exclusion Criteria:

* Present or previous diagnosis of any psychiatric disorder or major developmental disorder (autism/Asperger's disorder, pervasive developmental disorder), based on psychiatric evaluation using the Mini International Neuropsychiatric Interview (M.I.N.I.) or Structured Clinical Interview for DSM disorders (SCID)
* Any disability or health problem that prevents them from completing study procedures (e.g. color blindness, severe carpal tunnel syndrome, etc.)
* History of organic mental syndromes, head trauma, migraines, seizures, other CNS neurological disease, recent use of illegal drugs or current substance dependence, or significant medical illness other than that listed above (by self-report)
* Pregnant or nursing women
* Subjects with a medical condition or other predisposition that increases the risk of adverse effects when taking ondansetron. These include individuals with drug allergies or known hypersensitivity to ondansetron (or other 5-HT3 antagonists), heart disease, congestive heart failure, heart rhythm disorder, congenital long QT syndrome, electrolyte abnormalities (e.g., hypokalemia, hypomagnesemia) or hepatic impairment
* Subjects who report taking apomorphine will be excluded
* Subjects with abnormal EKG will either be excluded from participation, or referred to a cardiologist for further assessment of eligibility
* Subjects with abnormal liver function or electrolytes (as determined by blood test) will be excluded from participation if a study team physician determines it is unsafe for them to participate
* Cross-reactivity with other 5-HT3 antagonists has been reported, so any individual taking a 5-HT3 antagonist will be excluded

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2015-08; Primary Completion 2017-02-03 (Actual); Study Completion 2017-02-03 (Actual)

PRIMARY OUTCOMES:
BOLD signal in the insula and somatosensory cortex measured by fMRI | Day 1
  On Day1, Functional magnetic resonance imaging (fMRI) will be done 90 minutes after drug or placebo ingestion to measure the blood oxygen level dependent (BOLD) signal in insula and somatosensory cortex.
BOLD signal in the insula and somatosensory cortex measured by fMRI | 1 week
  At week 1, fMRI will be done 90 minutes after drug or placebo ingestion to measure the BOLD signal in insula and somatosensory cortex.

SECONDARY OUTCOMES:
BOLD signal in the whole brain measured by fMRI | Day 1
  On Day1, fMRI will be done 90 minutes after drug or placebo ingestion to measure the BOLD signal across the whole brain.
BOLD signal in the whole brain measured by fMRI | 1 week
  At week 1, fMRI will be done 90 minutes after drug or placebo ingestion to measure the BOLD signal across the whole brain.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Stern, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States